CLINICAL TRIAL: NCT01119417
Title: The Role of Endothelin in the Supine Hypertension of Autonomic Failure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 091344
Record Dates: First submitted 2010-05-04; First posted 2010-05-07 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Hypertension; Pure Autonomic Failure; Multiple System Atrophy
Keywords: supine Hypertension; autonomic failure; BQ123; BQ-123; endothelin
MeSH Terms: conditions — Hypertension; Pure Autonomic Failure; Multiple System Atrophy | interventions — cyclo(Trp-Asp-Pro-Val-Leu); Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BQ123 (Experimental): endothelin blocker
  Interventions: Drug: BQ123
- Saline (Placebo Comparator): IV saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: BQ123 — Low dose day: 25 nmol/min, single IV infusion for 15 min.
  Other Names: BQ-123 sodium salt
  Arms: BQ123
Drug: BQ123 — Low dose day: 50 nmol/min, single IV infusion for 15 min
  Other Names: BQ-123 sodium salt
  Arms: BQ123
Drug: Bq123 — High dose day: 100 nmol/min, single IV infusion for 15 min.
  Other Names: BQ-123 sodium salt
  Arms: BQ123
Drug: BQ123 — High dose day: 300 nmol/min, single IV infusion for 15 min.
  Other Names: BQ-123 sodium salt
  Arms: BQ123
Drug: Saline — 2-3 IV saline infusions for 15 min each.
  Other Names: Normal saline, 0.9% sodium chloride
  Arms: Saline

SUMMARY:
The purpose of this study is to test the hypothesis that endothelin plays a role in the pathogenesis of supine hypertension in pure autonomic failure by increasing vascular resistance. To gauge its contribution to blood pressure regulation, pure autonomic failure and multiple system atrophy patients with supine hypertension will undergo a medication testing with the endothelin blocker, BQ123. We will compare the hemodynamic effects between PAF and MSA patients. Our primary endpoint will be the decrease in blood pressure during the administration of this compound.

DETAILED DESCRIPTION:
The pathophysiologic mechanisms causing supine hypertension in patients with autonomic failure are not completely understood.In MSA patients, supine hypertension may be explained by residual sympathetic tone, possibly acting on hypersensitive adrenoreceptors and unstrained by the lack of baroreflex modulation. In contrast, the pathogenesis of hypertension in PAF remains unknown. Hypertension in these patients is not related to intravascular volume, residual sympathetic tone, or renin mechanisms. Increased vascular resistance is the underlying hemodynamic mechanism. The driving force of this increased vascular tone, however, is not known.

We hypothesize that endothelin (ET)-l contributes to the increased vascular resistance in pure autonomic failure patients with supine hypertension. To gauge its contribution to blood pressure regulation, we will induce endothelin blockade with acute systemic administration of BQ123 in an ascending dose regimen (25, 50, 100 and 300 nmol/min) and we will compare the hemodynamic effects between PAF and MSA patients.

Subjects will be studied on 3 different days, one with saline (placebo) and two with BQ123: a 'low dose' day (25 and 50 nmol/min infusions separated by 75 min) and a 'high dose' day (100 and 300 nmol/min infusions separated by 75 min). The order of the placebo day will be randomized in a single-blinded manner so that each subject receives it on a different visit. The order of the BQ123 study days will be always the same, starting with the low dose. If SBP drops by >40 mm Hg or SBP < 130 mm Hg during the monitoring period after the first or second infusion, the following dose(s) of BQ123 will not be given and patients will receive normal saline until the study ends.

Ganglionic Blockade with Trimethaphan (optional study day):

The purpose of this study day is to determine the level of residual sympathetic tone that contributes to supine hypertension in each autonomic failure patient by inducing transient withdrawal of the autonomic nervous system. This approach would allow us to identify patients in whom supine hypertension is not driven by sympathetic tone and thus, better characterize the role of endothelin in the hypertension of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with autonomic failure and supine hypertension from all races, who are in the hospital participating in the study "The Evaluation and Treatment of Autonomic Failure" (IRB# 000814).
* Supine hypertension, defined as a systolic blood pressure >150 mm Hg or diastolic blood pressure > 90 mm Hg.
* Males and females, between 18-85yr.
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care.

Exclusion Criteria:

* Pregnant women.
* High-risk patients (e.g. heart failure, symptomatic coronary artery disease, liver impairment, history of stroke or myocardial infarction).
* History of serious allergies or asthma.
* In the investigator's opinion, have clinically significant abnormalities on clinical, mental examination or laboratory testing.
* All medical students.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change in Systolic BP | 0 -4 hr post infusion
  Change from baseline in systolic blood pressure

SECONDARY OUTCOMES:
Change in cardiac output, stroke volume and systemic vascular resistance | 0-4 hr post infusion
  Percent change from baseline in hemodynamic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No